CLINICAL TRIAL: NCT02955901
Title: A 3-day Versus 1-day Low Residue Diet to Improve Colonoscopy Preparation Result and Patient Tolerability: A Prospective, Randomized, Single-blinded, Controlled Trial
Brief Title: 3-day vs. 1-day Low Residue Diet Influence in Colonoscopy Preparation and Patient Tolerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Filipe Taveira, Principal Investigator, Portuguese Oncology Institute, Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PortugueseOIC 002
Record Dates: First submitted 2016-10-25; First posted 2016-11-04 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Colon Disease; Colonic Neoplasms
Keywords: Randomized controlled trial; Colonoscopy; Colon Disease; Low residue diet; Colon preparation
MeSH Terms: conditions — Colonic Diseases; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-day low residue diet (Active Comparator): Group A - 3 day low residue diet prior to the colonoscopy
  Interventions: Other: 3 day low residue diet prior to the colonoscopy
- 1-day low residue diet (Placebo Comparator): Group B - 1 day low residue diet prior to the colonoscopy
  Interventions: Other: 1 day low residue diet prior to the colonoscopy

INTERVENTIONS:
Other: 3 day low residue diet prior to the colonoscopy — 3 day low residue diet prior to the colonoscopy
  Arms: 3-day low residue diet
Other: 1 day low residue diet prior to the colonoscopy — 3 day low residue diet prior to the colonoscopy
  Arms: 1-day low residue diet

SUMMARY:
Colonoscopy is one of the most common methods for the diagnosis and treatment of lower gastrointestinal tract diseases and provides a unique opportunity to identify early neoplastic lesions.

Adequate bowel preparation is important for optimal colonoscopy. New bowel-cleansing regimens, study of patient-related risk factors to fail a proper preparation and diet adaptations have been studied recently.

A low residue diet is the standard in the day before the colonoscopy. Some endoscopists prescribe this dietary plan for a 3-day period prior to the exam, although no study compared the recommended 1-day versus 3-day diet regime, or the influence in bowel preparation results.

The aim of this project is to determine if the use of a 3-day low residue diet improves bowel preparations results and the influence in patient tolerability and adherence.

DETAILED DESCRIPTION:
a. Study type: prospective, randomized, single-blinded trial:

i. Prospective inclusion of ambulatory patients;

ii. Randomization by computer generated tables;

iii. Allocation concealment by sealed, opaque envelopes;

iv. Patient not blinded to diet;

v. Endoscopist blinded to the diet followed by each patient.

b. Patient selection: Consecutive series of patients scheduled for total colonoscopy; Exclusion criteria: inpatients, sedation, urgent procedures, colonoscopies not intended to reach the caecum, patient with previous partial colectomy.

c. Sample Size:

i. 412 individuals; 2 groups of 206 patients

ii. Primary goal: to achieve a reduction from 15 to 5% of inappropriate preparation result; The Boston Bowel Preparation Scale (BBPS) will be used as grading system. Inappropriate is defined as total BBPS < 6 or < 2 in any segment. The chosen scale is the most systematically validated and appropriate for the clinical setting. iii.Both groups, from a community-based outpatient ambulatory center, used the same split dose regimen with Polyethylene glycol (PEG).Patients were instructed to drink 3 L of PEG preparation on the afternoon of the day prior to the exam and 1 L four hours before the scheduled exam time. All the exams scheduled for morning period. Assuming a normal distribution, a power of 90% and a type I error of 0.05, the calculated sample size for each group was 188; allowing a 10% dropout rate, the sample size is 206 per group (412 patients overall); Groups: Group A: 3-day low residue diet + split dose preparation; Group B: 1-day low residue diet + split dose preparation

d. Endoscopist:

Exams to be conduct by 5 board-certified gastroenterologists and 2 supervised fellows in training; All physicians were trained in the use of BBPS by online training available at http://cori.org/bbps/, and have been using the BBPS for at least 3 months.

e. Data collection methods: form sheet filled by the endoscopist and patient opinion regarding the assigned bowel preparation protocol.

f. Analyzed variables:

i. Primary outcome: BBPS score

ii. Secondary outcome: Patient assessment of tolerance and acceptance of the preparation and diet

iii. Tertiary outcome: polyp detection rate (PDR), polyp location, size and configuration; adenoma detection rate (ADR), cecum intubation rate

iv. Other variables and patients characteristics (age, gender, chronic medication, risk factors for inappropriate preparation), withdrawal time.

g. Statistical analysis: T-test for groups comparing quantitative variables with normal distribution (primary outcome); Qui square test for groups comparing proportions (secondary and tertiary outcomes)

ELIGIBILITY:
Inclusion Criteria:

* Consecutive series of patients scheduled for total colonoscopy
* Signed informed consent

Exclusion Criteria:

* inpatients
* sedation
* urgent procedures
* colonoscopies not intended to reach the caecum
* patient with previous partial colectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Score of mucosal visualization | 1 day (during colonoscopy)
  Using Boston Bowel Preparation Scale during the exam

SECONDARY OUTCOMES:
Patient assessment of diet protocol | 1 day (the day of the exam)
  Patient assessment, by written questionnaire, of tolerance and acceptance of diet protocol.
Polyp detection rate, location and configuration | 1 day (during colonoscopy)
  One of the quality indicators for colonoscopy is polyp detection rate, which is defined as the percentage of colonoscopies with a detection of at least one polyp. At the same time the endoscopist will assign the colonic location of the polyp (ascendent, transverse, descendent).
  (PDR to be presented as %; Location to be discriminated in the endoscopist report).
Adenoma Detection Rate | Within 30 days from colonoscopy date
  Adenoma detection rate (ADR) is the one of the strongest quality indicators for colonoscopy. This rate represents the percentage of colonoscopies with at least one adenoma identified. (to be presented as %)
Cecum intubation rate | 1 day (during colonoscopy)
  Defined as colonoscopy quality indicator the photo documentation of cecum, in at least 95% of the colonoscopies. Photo documentation of the cecum is a mark for effective total colonoscopy. (to presented as %)
Withdrawal time | 1 day (during colonoscopy)
  In a negative colonoscopy (no polyp identification) is defined that the withdrawal time should be at least 6 minutes for proper and safe colonic mucosa evaluation. (to be presented in minutes)

OTHER OUTCOMES:
Patients characteristics questionnaire | 1 day
  Evaluate, using proper data collecting sheet, patient relevant data (age, gender, chronic medication, risk factors for inappropriate preparation)

CONTACTS AND LOCATIONS:
Overall Officials: Filipe Taveira, MD, Principal Investigator — Portuguese Oncology Institute, Coimbra
Locations (1):
- Portuguese Oncology Institute - Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Gastrointest Endosc. 2015 Jan;81(1):31-53. doi: 10.1016/j.gie.2014.07.058. Epub 2014 Dec 2. No abstract available. PMID 25480100
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] Bucci C, Rotondano G, Hassan C, Rea M, Bianco MA, Cipolletta L, Ciacci C, Marmo R. Optimal bowel cleansing for colonoscopy: split the dose! A series of meta-analyses of controlled studies. Gastrointest Endosc. 2014 Oct;80(4):566-576.e2. doi: 10.1016/j.gie.2014.05.320. Epub 2014 Jul 19. PMID 25053529
- [Background] Cohen LB. Advances in bowel preparation for colonoscopy. Gastrointest Endosc Clin N Am. 2015 Apr;25(2):183-97. doi: 10.1016/j.giec.2014.11.003. Epub 2015 Jan 9. PMID 25839681
- [Background] Hautefeuille G, Lapuelle J, Chaussade S, Ponchon T, Molard BR, Coulom P, Laugier R, Henri F, Cadiot G. Factors related to bowel cleansing failure before colonoscopy: Results of the PACOME study. United European Gastroenterol J. 2014 Feb;2(1):22-9. doi: 10.1177/2050640613518200. PMID 24918005
- [Background] Song GM, Tian X, Ma L, Yi LJ, Shuai T, Zeng Z, Zeng XT. Regime for Bowel Preparation in Patients Scheduled to Colonoscopy: Low-Residue Diet or Clear Liquid Diet? Evidence From Systematic Review With Power Analysis. Medicine (Baltimore). 2016 Jan;95(1):e2432. doi: 10.1097/MD.0000000000002432. PMID 26735547
- [Background] Nguyen DL, Jamal MM, Nguyen ET, Puli SR, Bechtold ML. Low-residue versus clear liquid diet before colonoscopy: a meta-analysis of randomized, controlled trials. Gastrointest Endosc. 2016 Mar;83(3):499-507.e1. doi: 10.1016/j.gie.2015.09.045. Epub 2015 Oct 13. PMID 26460222
- [Background] Lijoi D, Ferrero S, Mistrangelo E, Casa ID, Crosa M, Remorgida V, Alessandri F. Bowel preparation before laparoscopic gynaecological surgery in benign conditions using a 1-week low fibre diet: a surgeon blind, randomized and controlled trial. Arch Gynecol Obstet. 2009 Nov;280(5):713-8. doi: 10.1007/s00404-009-0986-3. Epub 2009 Feb 20. PMID 19229545
- [Background] Vanhauwaert E, Matthys C, Verdonck L, De Preter V. Low-residue and low-fiber diets in gastrointestinal disease management. Adv Nutr. 2015 Nov 13;6(6):820-7. doi: 10.3945/an.115.009688. Print 2015 Nov. PMID 26567203
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Parmar R, Martel M, Rostom A, Barkun AN. Validated Scales for Colon Cleansing: A Systematic Review. Am J Gastroenterol. 2016 Feb;111(2):197-204; quiz 205. doi: 10.1038/ajg.2015.417. Epub 2016 Jan 19. PMID 26782820
- See also: BBPS training — http://cori.org/bbps/